CLINICAL TRIAL: NCT06396962
Title: Survival and Prognostic Factors of Primary Retroperitoneal Sarcomas After Surgery: a Single-center Experience
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Dr, Northern Jiangsu People's Hospital
Other Study IDs: Northjiangsu010
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Primary Retroperitoneal Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: WANG DAORONG — surgery

SUMMARY:
he percentage of retroperitoneal sarcomas (RPS) among all soft tissue sarcomas ranges from 10%-15%. Surgery remains the gold standard for RPS. In this study, we analyzed the impact of surgical treatment for primary RPS on recurrence and overall mortality at a Chinese institution and identified and evaluated prognostic variables.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were as follows: (1) diagnosis of primary retroperitoneal sarcoma, (2) pathological conformity, (3) no prior surgical resection, (4) complete clinicopathological data, and (5) age of ≥18.

Exclusion Criteria:

* Patients with benign retroperitoneal tumors, gastrointestinal stromal tumors, Ewing, desmoid-type fibromatosis, pheochromocytomas/paragangliomas, or any other subtypes other than RPS were not included. The ethics committee of the Northern Jiangsu People's Hospital approved the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: (1) diagnosis of primary retroperitoneal sarcoma, (2) pathological conformity, (3) no prior surgical resection, (4) complete clinicopathological data, and (5) age of ≥18.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No